CLINICAL TRIAL: NCT04112641
Title: Alleviation by NIAGEN of Persistent Chemotherapy-Induced Peripheral Neuropathy in Cancer Survivors
Brief Title: NIAGEN and Persistent Chemotherapy-Induced Peripheral Neuropathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Donna Hammond, PhD (Other)
Responsible Party: Sponsor-Investigator, Donna Hammond, PhD, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201909843
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: peripheral neuropathy; chemotherapy; taxane; platinum compound
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Two independent treatment arms to which patients will be randomized by variable size blocks
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Placebo capsules and drug capsules look alike
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo capsules (Placebo Comparator): Subjects will take 2 capsules in the a.m. and 2 capsules in the p.m. daily for 84 days.
  Interventions: Drug: Placebo capsules
- Nicotinamide Riboside (NIAGEN) (Experimental): Subjects will take 2 250-mg capsules in the a.m. and 2 250- mg capsules in the p.m. daily (total daily dose is 1 g) for 84 days.
  Interventions: Drug: Nicotinamide riboside

INTERVENTIONS:
Drug: Nicotinamide riboside — Daily oral ingestion of 1 g/day NIAGEN in capsule form for 84 days; two capsules in the a.m. and two capsules in the p.m.
  Other Names: NIAGEN
  Arms: Nicotinamide Riboside (NIAGEN)
Drug: Placebo capsules — Daily oral ingestion of placebo in capsule form for 84 days; two capsules in the a.m. and two capsules in the p.m.
  Other Names: Placebo
  Arms: Placebo capsules

SUMMARY:
The purpose of this randomized, double-blind, placebo-controlled, parallel group phase II trial is to determine whether nicotinamide riboside (NIAGEN®, NR) can ameliorate persistent peripheral neuropathy in cancer survivors who have completed chemotherapy with taxane or platinum-complex compounds between 1 and 12 months earlier.

DETAILED DESCRIPTION:
Patients who have been declared to be in complete remission after treatment of their cancer with either taxane or platinum-based compounds and who have persistent neuropathy will be randomized to receive either placebo or NIAGEN capsules daily for 84 days. On enrollment, subjects will complete several questionnaires characterizing the type and severity of their neuropathy. Their fifth finger will be scanned to determine the density of sensory afferents in the skin, and a skin biopsy will be taken above the ankle for histological analysis of nerve fiber density. Blood samples will be drawn for baseline measures of NAD+ levels, and clinical chemistries and indices of liver and kidney function. Subjects will be asked to return every two weeks to complete the questionnaires, and blood will be drawn to measure biomarkers of NIAGEN consumption. Blood will be drawn at visits on days 28, 56, and 84 for clinical chemistries and measures of liver and kidney function. At visits on day 42 and 84, additional measures of density of nerve fibers in the hand and leg will be made. The last treatment day will be day 84, at which time all measures will be redetermined. A follow-up period of 3 months is planned at which time all measures will be conducted once again to determine if any alleviation of the chemotherapy has persisted after treatment ended. Patients enrolled in this study will receive standard of care treatment by their oncologists, which includes computed tomography, magnetic resonance or ultrasound scans every three months as surveillance for cancer re-occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent and HIPAA authorization
* Be ≥ 18 and ≤ 85 years of age
* Have received chemotherapy with taxane (e.g. paclitaxel, nab-paclitaxel, or docetaxol) or platinum-complex (e.g. oxaliplatin, carboplatin, or cisplatin) (alone or in combination) and completed therapy no sooner than 1 month and no later than 1 year earlier.
* Have been treated with above compounds for head and neck cancer, small cell lung cancer, sarcoma, ovarian cancer, endometrial cancer, colorectal cancer, or breast cancer and been declared to have no visible evidence of disease.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Able to take medication orally - up to four capsules in the morning (am) and four capsules in the evening (pm).
* Be determined to have a raw score of ≥ 12 on the sensory subscale or ≥ 11 on the motor subscale of the QLQ-CIPN20 questionnaire.
* Females must be either postmenopausal for at least 1 year or surgically sterile for at least 6 weeks. Females of childbearing potential must have a negative pregnancy test at screening to be eligible for study participation and agree to take appropriate precautions to avoid pregnancy from screening through follow-up.
* Males must agree to take appropriate precautions to avoid fathering a child from screening through follow-up. The following methods have been determined to be more than 99% effective (<1% failure rate per year when used consistently and correctly) [69] and are permitted under this protocol for use by the patient and his/her partner:

  * Complete abstinence from sexual intercourse when this is in line with the preferred and usual lifestyle of the patient
  * Double barrier methods
  * Condom with spermicide in conjunction with use of an intrauterine device
  * Condom with spermicide in conjunction with use of a diaphragm
  * Surgical sterilization (bilateral oophorectomy with or without hysterectomy, tubal ligation or vasectomy) at least 6 weeks prior to taking study treatment. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up levels of luteinizing hormone (LH), follicle-stimulating hormone (FSH), and/or estradiol
  * Non-hormonal intrauterine device used as directed by provider placing this is also acceptable.

Exclusion Criteria:

* Pre-existent peripheral neuropathy that is unrelated to chemotherapy
* Recurrent ovarian or endometrial cancer
* Diabetes managed by medication
* Neutrophils < 1,000 cells/m3
* Hemoglobin < 8.0 g/dcl
* Platelets < 100,000 cells/m3
* Creatinine clearance < 30 ml/min
* aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values > 2.5 X upper limits of normal
* Total bilirubin > 2.0 X upper limits of normal
* Heavy alcohol use defined at > 8 drinks/week by women or 12 drinks/week by men
* Psychiatric illness that, in the opinion of the investigator, would interfere with the ability of the individual to participate in or complete the study.
* Pregnancy
* Current imprisonment
* Limitations of self-expression, defined as an inability to answer questions posed by physicians, nurses, care-givers, or other members of the investigative team or an inability to describe somatosensations.
* Known HIV
* Regular use of nutritional supplements that contain nicotinamide riboside (e.g. NIAGEN, TRuNIAGEN, Basis, NAD+ Cell Regenerator) within the previous 30 days
* Use of duloxetine (Cymbalta®) or any other drug for treatment of peripheral neuropathy such as gabapentin, pregabalin, lamotrigine, or amitryptyline.
* Pancreatic insufficiency requiring exocrine enzyme replacement therapy
* GI conditions where malabsorption of B complex vitamins is known to occur.
* Breastfeeding
* Allergy to epinephrine or local anesthetics
* Bleeding disorder

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Score on Sensory Subscale of Quality of Life Questionnaire Chemotherapy-induced Peripheral Neuropathy (QLQ-CIPN20) | 84 days
  Change in score from baseline to end of treatment at 84 days. The Quality of Life Questionnaire for Chemotherapy-induced Peripheral Neuropathy (20 questions) or QLQ-CIPN20 yields scores of 1-4 (Likert scale) for 9 sensory, 8 motor, and 3 autonomic sequelae of chemotherapy. The minimum score for the sensory subscale is 9 and the maximum possible score is 36. The higher the score, the worse the signs and symptoms. The raw score can, at the investigator's discretion, be linearly transformed to a 0-100 scale, where higher numbers represent worse symptoms.
  Recent publications call the validity of the autonomic scale into question, and it is not being used in this study.
Score on Motor Subscale of Quality of Life Questionnaire Chemotherapy-induced Peripheral Neuropathy (QLQ-CIPN20) | 84 days
  Change in score from baseline to end of treatment at 84 days. The Quality of Life Questionnaire for Chemotherapy-induced Peripheral Neuropathy (20 questions) or QLQ-CIPN20 yields scores of 1-4 (Likert scale) for 9 sensory, 8 motor, and 3 autonomic sequelae of chemotherapy. The minimum score for the motor subscale is 8 and the maximum possible score is 32. The higher the score, the worse the signs and symptoms. The raw score can, at the investigator's discretion, be linearly transformed to a 0-100 scale, where higher numbers represent worse symptoms.
  Recent publications call the validity of the autonomic scale into question, and it is not being used in this study.

SECONDARY OUTCOMES:
Total Neuropathy Score - clinical questionnaire | 84 days
  Change in score from baseline to end of treatment at 84 days. The clinical version of the Total Neuropathy Score yields scores of 0-4 on 6 items (sensory symptoms, motor symptoms, pin sensibility, vibration sensibility, strength and deep tendon reflex). The minimum possible score is 0 and the maximum possible score is 30. Scores for each of the six items are summed to yield a single total score. The higher the score, the worse the outcome.
Intraepidermal Nerve Fiber Density | 84 days
  Change in score from baseline to end of treatment at 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Milhem, M.D., Principal Investigator — University of Iowa; Donna Hammond, Ph.D., Principal Investigator — University of Iowa; Michael Shy, M.D., Principal Investigator — University of Iowa
Locations (1):
- Donna Hammond, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No